CLINICAL TRIAL: NCT01892813
Title: Tailored Tobacco Intervention
Brief Title: Dissemination of a Tailored Tobacco Quitline for Rural Veteran Smokers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mark Vander Weg (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mark Vander Weg, Associate Professor of Internal Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201305740
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Nicotine Dependence; Tobacco Use
Keywords: Nicotine dependence; Smoking cessation; Telehealth; Alcohol use; Depression; Body weight
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Smoking Cessation; Alcohol Drinking; Depression; Body Weight | interventions — Bupropion; Varenicline; Nicotine Chewing Gum; Tobacco Use Cessation Devices; Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored intervention (Experimental): Participants will receive a combined behavioral and pharmacological intervention. The behavioral component will consist of a six-session cognitive behavioral telephone intervention combined with supplemental treatment modules to address common issues (symptoms of depression, weight gain, risky alcohol use) associated with cigarette smoking based on eligibility and preference.
  Interventions: Drug: Nicotine replacement therapy - Transdermal nicotine patch; Drug: Nicotine replacement therapy - Nicotine gum; Drug: Nicotine replacement therapy - Nicotine lozenge; Drug: Bupropion; Drug: Varenicline; Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine gum; Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine lozenge; Drug: Combination pharmacotherapy - Transdermal nicotine patch + bupropion; Behavioral: Tailored behavioral intervention; Behavioral: Alcohol use risk reduction; Behavioral: Behavioral activation for depressive symptoms; Behavioral: Behavioral management of postcessation weight gain
- Enhanced standard of care (Active Comparator): Participants assigned to the enhanced standard of care condition will receive referral to their state tobacco quitline along with pharmacotherapy to assist with smoking cessation.
  Interventions: Drug: Nicotine replacement therapy - Transdermal nicotine patch; Drug: Nicotine replacement therapy - Nicotine gum; Drug: Nicotine replacement therapy - Nicotine lozenge; Drug: Bupropion; Drug: Varenicline; Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine gum; Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine lozenge; Drug: Combination pharmacotherapy - Transdermal nicotine patch + bupropion; Behavioral: Tobacco quitline referral

INTERVENTIONS:
Drug: Nicotine replacement therapy - Transdermal nicotine patch — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
Drug: Nicotine replacement therapy - Nicotine gum — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
  Other Names: Nicotine polacrilix
Drug: Nicotine replacement therapy - Nicotine lozenge — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
  Other Names: Nicotine polacrilix
Drug: Bupropion — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
  Other Names: Zyban
Drug: Varenicline — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
  Other Names: Chantix
Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine gum — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
Drug: Combination pharmacotherapy - Transdermal nicotine patch + nicotine lozenge — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
Drug: Combination pharmacotherapy - Transdermal nicotine patch + bupropion — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
Behavioral: Tobacco quitline referral — Participants assigned to this condition will receive a referral to their state tobacco quitline. The specific behavioral treatment that is provided will differ slightly depending upon the services available through the participant's state of residence.
  Arms: Enhanced standard of care
Behavioral: Tailored behavioral intervention — Participants will receive a standard six session cognitive behavioral intervention for smoking cessation combined with supplemental treatment modules based on individual need and preference.
  Arms: Tailored intervention
Behavioral: Alcohol use risk reduction — Participants engaging in risky alcohol use may receive this six-session telephone-based behavioral intervention for reducing alcohol use.
  Other Names: Harm reduction
  Arms: Tailored intervention
Behavioral: Behavioral activation for depressive symptoms — Participants with elevated depressive symptoms may receive this six-session telephone-based behavioral activation intervention.
  Arms: Tailored intervention
Behavioral: Behavioral management of postcessation weight gain — Participants with concerns about gaining weight after quitting smoking may receive this six-session telephone-based behavioral self-management intervention designed to help attenuate post-cessation weight gain.
  Other Names: Weight management
  Arms: Tailored intervention

SUMMARY:
The project is designed to examine the effectiveness of strategies to increase access to treatment for tobacco use and dependence among rural Veteran smokers. In addition, it will examine whether tailored treatment that is designed to address common comorbid conditions that are related to cigarette smoking enhances success with quitting relative to enhanced standard of care. The investigators hypothesize that participants assigned to the tailored tobacco cessation intervention will report greater cessation rates at six months. The investigators also anticipate more favorable outcomes on measures of depressive symptoms, alcohol use, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* 18 + years of age
* Smoke cigarettes on at least a daily basis
* Receive primary care from the Iowa City VA Health Care System or an affiliated Community-based Outpatient Clinic (CBOC)
* Live in a non-metropolitan area (based on Rural-Urban Commuting Area Codes (RUCA) codes)
* Be willing to make an attempt to quit smoking in the next 30 days
* Be capable of providing informed consent
* Have access to a telephone (land line or cell phone)
* Have a stable residence

Exclusion Criteria:

* Planning to move within the next 12 months
* Presence of a terminal illness
* Pregnancy
* Unstable psychiatric disorder (e.g., acute psychosis)
* Currently pregnant
* Incarcerated
* Institutionalized

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2013-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Tobacco use | Six-month follow-up
  At the six-month follow-up contact, participants will be questioned regarding self-reported tobacco use over the past seven and 30 days.

SECONDARY OUTCOMES:
Alcohol use | Six-month follow-up
  Alcohol use during the previous seven days will be assessed at the six month follow-up. Based on this information, several metrics of alcohol consumption will be obtained including: 1) average number of drinking days per week, 2) average number of drinks per drinking day, 3) number of drinks per week 4) number of heavy drinking days, and 5) maximum drinks consumed on a single occasion.
Depressive symptoms | Six-month follow-up
  Depressive symptoms will be assessed at the six-month follow-up using the Patient Health Questionnaire 9 (PHQ-9).
Body weight | Six-month follow-up
  Change in body weight will be assessed via self-report and chart review at the six-month follow-up.
Physical Activity | Six-month follow-up
  Physical activity will be assessed by self-report at the six-month follow-up visit using the Rapid Assessment of Physical Activity (RAPA).
Dietary intake | Six-month follow-up
  Self-reported dietary intake will be measured at six months using the Starting the Conversation - Diet questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Vander Weg, Ph.D., Principal Investigator — VRHRC-CR
Locations (1):
- Iowa City VA Healthcare System, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273